CLINICAL TRIAL: NCT03731494
Title: Quality of Life Assessment Before and After Hyposensitization Treatment in Systemic Nickel Allergy Syndrome
Brief Title: Quality of Life in Systemic Nickel Allergy Syndrome
Status: Completed | Type: Observational
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Eleonora Nucera, Prof., Catholic University of the Sacred Heart
Other Study IDs: 1377/15 (13939/14)
Record Dates: First submitted 2018-11-02; First posted 2018-11-06 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Systemic Nickel Allergy Syndrome; Quality of Life
Keywords: Nickel allergy; Systemic nickel allergy syndrome; Health-related quality of life; Nickel oral hyposensitizing treatment; Diet; Short-Form 36-Item Health Survey; Psychological General Well Being Index; Minnesota Multiphasic Personality Inventory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nickel oral hyposensitization treatment: The patients take capsules at different doses in nickel content until reaching the maximum dose of 1.5 mcg per week for a total of 12 months.
  Interventions: Biological: Nickel oral hyposensitization treatment

INTERVENTIONS:
Biological: Nickel oral hyposensitization treatment — Nickel oral hyposensitization treatment (NiOHT) was performed with hard gelatin capsules containing Nickel sulphate (NiSO4) at different dosages (0.1 ng, 1 ng, 10 ng, 0.1 μg, 0.5 μg) and microcrystalline cellulose as excipient (TIO Nickel, Lofarma SpA, Milan, Italy). Treatment was given 3 times a week increasing progressively the dose from 0.1 ng to 3 μg in 10 weeks with a maintenance phase of 1,5 μg a week for a period of 12 months. After 6 months, patients were allowed to gradually reintroduce nickel-rich foods, starting with those with a maximum of 100 mcg of nickel content. For all the treatment period, information on the appearance of side effects or more severe adverse reactions and the need for antiallergic drugs (corticosteroids, antihistamine drugs) were collected.
  Other Names: NiOHT - TIO Nickel

SUMMARY:
This study evaluates the effects of Nickel oral hyposensitization treatment (NiOHT) on health-related quality of life (HRQoL) of patients suffered from Systemic Nickel Allergy Syndrome (SNAS).

DETAILED DESCRIPTION:
Nickel (Ni) is a nutritionally essential metal widely distributed in the environment, and it has been reported to be one of the most common causes of allergic contact dermatitis (ACD), affecting nearly 15-20% of the general population. As known, Ni-hypersensitivity can induce less frequently also respiratory allergy (RA) and in approximately 20% of Ni-ACD patients cause a more complex condition termed Systemic Nickel Allergy Syndrome (SNAS). It is characterized by a combination of cutaneous (in regions without direct nickel contact) and extracutaneous gastrointestinal symptoms, after the ingestion of Ni-rich foods, especially vegetables. Then, a low-Ni diet, following positive patch tests, represents a effective diagnostic and therapeutic tool in the control of systemic manifestations, determining a significant clinical improvement.

It is known that Nickel oral hyposensitization treatment (NiOHT) is a effective approach for the management of Ni allergy, especially in a subset of patients with SNAS, inducing immunological and clinical tolerance to metal at the doses normally taken with the diet.

Although a large number of clinical trials focused on the health-related quality of life (HRQoL) in allergic disease, the expectations, the needs and the psychosocial characteristics of patients affected by SNAS are limited and no data exist pre- and post-treatment and specifically with NiOHT. Given the high safety profile and beneficial effects of immunotherapy on HRQoL of patients with allergic rhinitis, we hypothesized similar positive results even after oral Ni desensitization.

ELIGIBILITY:
Inclusion Criteria:

* history of SNAS (coexistence of typical cutaneous and gastrointestinal symptoms),
* positive Ni-patch test,
* clinical improvement at least 70% from baseline after 4 weeks on a low-Ni diet,
* positivity of a double blind placebo-controlled oral Ni challenge (DBPCO),
* written informed consent.

Exclusion Criteria:

* age < 18 years and > 65 years,
* other organic gastrointestinal diseases, such as peptic ulcer, inflammatory bowel diseases, celiac disease, gastrointestinal infections, and small intestinal bacterial overgrowth,
* diabetes mellitus,
* hepatic, renal or cardiac dysfunction,
* thyroid disease or tumor,
* concomitant treatment with steroids and/or antihistamines in the previous 4 weeks, pregnancy, lactation,
* smoking, abuse of alcohol, coffee, tea, and cola intake,
* refusal to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Researchers enrol patients suffer from Systemic Nickel Allergy Syndrome (SNAS), condition characterised by a combination of cutaneous (in regions without direct nickel contact) and extracutaneous gastrointestinal symptoms, after the ingestion of Nickel-rich foods, especially vegetables.
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
QoL: Short-Form 36-Item Health Survey (SF-36v2) | Change from baseline index at 12 months
  Short-Form 36-Item Health Survey (SF-36v2) is a self-administered questionnaire comprising 36-items measuring eight dimensions of general HRQOL: physical functioning (10 items), role limitation due to physical health problems (4 items), bodily pain (2 items), general health perceptions (5 items), vitality (4 items), social functioning (2 items), role limitations due to emotional problems (3 items), and general mental health (5 items). In addition to scores for individual dimensions, two summary scores assessing physical and mental dimensions of health and well-being can also be calculated: Physical Component Summary (PCS) score and the Mental Component Summary (MCS) score, respectively.
QoL: Psychological General Well Being Index (PGWBI) | Change from baseline index at 12 months
  The PGWBI consists of 22 questions, which deal with six factors (anxiety, depression, vitality, general health,self-control and well-being) constituting a global assessment.The response format is graded 1-6 (i.e. total range 22-132), with the highest value corresponding to optimal well-being.

SECONDARY OUTCOMES:
Psychological state: Minnesota Multiphasic Personality Inventory (MMPI-2) | Baseline.
  The MMPI-2 questionnaire containing 567 items with 2 choices of answer ("true" or "false") in order to assess the main structural features of personality and emotional disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Eleonora Nucera, MD,Prof, Principal Investigator — Catholic University of Sacred Heart; Antonio Gasbarrini, MD,Prof, Study Director — Catholic University of Sacred Heart
Locations (1):
- Catholic University of Sacred Heart, Roma, Italy

IPD SHARING:
Plan to Share IPD: No